CLINICAL TRIAL: NCT05265975
Title: A Single-arm, Phase Ⅰ/Ⅱ Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of ATG-010 in Combination With Lenalidomide and Rituximab (R2) in Adult Patients With Relapsed/Refractory DLBCL and iNHL Who Are Ineligible for High-dose Chemotherapy (HDC) or Autologous Stem Cell Transplant (ASCT)
Brief Title: A Study of ATG-010 in Combination With Lenalidomide and Rituximab (R2) in Adults With DLBCL and iNHL
Acronym: SWATCH
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The adjustment of the sponsor's research and development strategy
Sponsor: Antengene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-010-B-NHL-002
Record Dates: First submitted 2022-02-09; First posted 2022-03-04 (Actual); Last update posted 2025-06-09 (Actual); Status verified 2025-03

CONDITIONS: Diffuse Large B-cell Lymphoma; Indolent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — selinexor; Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATG-010 (Experimental): Enrolled patients will be treated with dosage groups. Dosage group 1:40mg/time, dosage group 2:60mg/time, dosage group 3:80mg/time; The treatment period was 28 days. The drug was administered on day 1,8 and 15 of each cycle
  Interventions: Drug: ATG-010; Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: ATG-010 — Tablets,20mg, once a week: dosage group 1:40mg/time, dosage group 2:60mg/time, dosage group 3:80mg/time The treatment period was 28 days. The drug was administered on day 1,8 and 15 of each cycle
  Other Names: Selinexor
Drug: Lenalidomide — Oral administration,QD, Days 1-21 of each cycle
Drug: Rituximab — Intravenous injection Days 1 of each cycle, Cycles 1-6

SUMMARY:
A Single-arm, Phase Ⅰ/Ⅱ Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of ATG-010 in Combination with Lenalidomide and Rituximab (R2) in Adult Patients with Relapsed/Refractory DLBCL and iNHL Who are Ineligible for High-dose Chemotherapy (HDC) or Autologous Stem Cell Transplant (A SCT).

DETAILED DESCRIPTION:
A Single-arm, Phase Ⅰ/Ⅱ Study Evaluating the Safety, Tolerability, and Preliminary Efficacy of ATG-010 in Combination with Lenalidomide and Rituximab (R2) in Adult Patients with Relapsed/Refractory DLBCL and iNHL Who are Ineligible for High-dose Chemotherapy (HDC) or Autologous Stem Cell Transplant (ASCT).About 84 subjects are scheduled to be enrolled in the study,Maximum 24 (Dose Escalation Phase) and 60 (Dose Expansion Phase).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Pathologically confirmed DLBCL (including de novo DLBCL or DLBCL transformed from previously diagnosed indolent lymphoma [e.g., follicular lymphoma]) or B-cell iNHL with histological subtype limited to FL Grade 1, Grade 2, or Grade 3a or nodal or extranodal marginal zone lymphoma (MZL), based on criteria established by the World Health Organization (WHO) 2016 classification.
3. Received at least 1 line of systemic therapy for the treatment of B-NHL.
4. Have evidence of relapse or refractory disease.
5. At least one bi-dimensionally measurable lesion per the Lugano 2014 Criteria (Cheson, 2014; Appendix 4).
6. Adequate bone marrow function at screening, defined as:

(1) absolute neutrophil count (ANC) ≥1.0 × 109/L (without hematopoietic stimulators such as granulocyte or granulocyte-macrophage colony stimulating factor within 7 days prior to testing); (2) Platelet count ≥75 × 109/L; or ≥50 × 109/L when lymphoma infiltrates bone marrow (without platelet transfusion or TPO, IL-11 and other hematopoietic stimulating factors administration within 7 days prior to testing); (3) Hemoglobin ≥80 g/L (without red blood cell transfusion or hematopoietic stimulating factor such as TPO administration within 14 days prior to testing).

7. Adequate liver and kidney function, defined as:

1. Aspartate transaminase (AST) or alanine transaminase (ALT) ≤2.5 × upper limit of normal (ULN);
2. Serum total bilirubin ≤1.5 × ULN, or ≤3 ULN if have Gilbert syndrome;
3. Calculated creatinine clearance (CrCl) ≥60 mL/min for Dose Escalation Phase, and ≥30 mL/min for Dose Expansion Phase, based on Cockcroft-Gault formula.

8. Eastern Cooperative Oncology Group (ECOG) performance status of ≤2. 9. Agree to effective contraception during the study and within 12 months after the last dose of study treatment.

Exclusion Criteria:

1. DLBCL with MALT lymphoma; composite lymphoma (Hodgkin's lymphoma+NHL); primary mediastinal (thymic) large B-cell lymphoma; Grade 3b follicular lymphoma.
2. Dose Escalation Phase: Subjects with known central nervous system involvement. Dose Expansion Phanse: Subjects with advanced lymphoma of the central nervous system involvement at screening, however, subjects have stable central nervous system lymphoma (in the case of no intracranial pressure or other conditions need medical intervention) or do not occur disease progression as assessed by neurological symptoms, signs, and radiography within 28 days prior to C1D1, will be considered eligible.
3. Previous treatment with ATG-010 (selinexor) or other XPO1 inhibitors, or prior exposure to lenalidomide within 3 months before C1D1.
4. Contraindication to any drug in the combination therapy of SR2.
5. Use of any standard or experimental anti B-NHL therapy <21 days prior to C1D1, including chemotherapy, immunotherapy, radio-immunotherapy, nonpalliative radiation, or any other anticancer therapy.
6. Major surgery, or live vaccines received <28 days prior to C1D1.
7. ASCT <6 months or CAR-T cell infusion <6 months prior to the screening.
8. History of allogeneic hematopoietic stem cell transplant.
9. Any AE related with prior B-NHL treatment had not recovered to ≤Grade 1 (CTCAE, v5.0) or baseline at Screening (except alopecia, AE related to hematology and blood biochemistry; the values of hematology and biochemistry refer to inclusion criteria 7 and 8).
10. Have active hepatitis B virus (HBV), hepatitis C virus (HCV) infections at screening.
11. Known serum HIV antibody positive or history of active HIV infection.
12. Active infection requiring intravenous antibiotics, antivirals, or antifungals treatment within 14 days prior to C1D1; however, prophylactic use of these agents is acceptable (including intravenous medication).
13. Prior malignancy that required treatment or has shown evidence of recurrence (except for non-melanoma skin cancer or adequately treated cervical carcinoma in situ) within the 2 years prior to C1D1.
14. Ischemic or hemorrhagic cerebrovascular disease, or gastrointestinal hemorrhage ≥Grade 3 (CTCAE, v5.0) within 6 months prior to screening.
15. History of deep vein thrombosis or pulmonary embolism within 12 months prior to screening.
16. Inability to swallow tablets, malabsorption syndrome, or any other gastrointestinal disease or dysfunction that could interfere with absorption of study treatment.
17. Inability or unwillingness to sign an ICF.
18. Existed any life-threatening illness, medical condition, or organ system dysfunction which, in the Investigator's opinion, could compromise the subject's safety, or being compliant with the study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
DLT | 28 days after administration
  The occurrence of severe toxicities during the first cycle of systemic cancer therapy
AE | 28 days after administration
  Any adverse medical event that occurs after a patient or clinical trial subject receives a drug product, but is not necessarily related to the treatment.

SECONDARY OUTCOMES:
ORR | One year after last patient first dose
  Percentage of subjects with PR, or CR
PFS | One year after last patient first dose
  Duration of time from the first dose of study drug until progression or death due to any cause
DOR | One year after last patient first dose
  Duration of time from first occurrence of CR or PR until the first date that disease
OS | One year after last patient first dose
  Duration of time from the first dose of study drug until death due to any cause

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The Second Affiliated Hospital of PLA Army Medical University, Chongqing, Chongqing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - The first Affiliated Hospital of China medical University, Shenyang, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality